CLINICAL TRIAL: NCT00894023
Title: IntraCoronary Abciximab With the ClearWay Catheter To Improve Outcomes With Lysis
Brief Title: Intracoronary Abciximab With Clearway Catheter
Acronym: IC-CLEARLY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the study was stopped because the sample size was very difficult to achieve.
Sponsor: Gennaro Sardella (Other)
Responsible Party: Sponsor-Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARD03
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Patients with AMI
MeSH Terms: interventions — Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abciximab (Experimental): IC bolus of abciximab
  Interventions: Drug: Intracoronary bolus wtih ClearWay™RX catheter
- IV Abciximab (Active Comparator): IV abciximab + infusion
  Interventions: Drug: IV abciximab

INTERVENTIONS:
Drug: Intracoronary bolus wtih ClearWay™RX catheter — Intracoronary bolus with Clearway catheter
  Arms: Abciximab
Drug: IV abciximab — IV abciximab + infusion
  Arms: IV Abciximab

SUMMARY:
Background: Percutaneous coronary intervention (PCI) is a highly effective therapy for acute ST-elevation myocardial infarction (STEMI). Adjunctive therapy with glycoprotein (GP) IIb/IIIa inhibitor can result in increased patency and improved outcomes in STEMI patients, with thrombus, undergoing PCI. The investigation of novel dosing and delivery strategies of this therapy may help to further improve outcomes.

Study design: Intracoronary Abciximab With Clearway Catheter trial is a randomized, open-label, multicenter, trial to evaluate the effect of an intracoronary (IC) bolus dose of abciximab delivered using the ClearWay™RX catheter versus an intravenous bolus (IV) of abciximab for STEMI with angiographically visible thrombus (Thrombus Grade > 2). All patients in both arms will receive intravenous abciximab infusion following the PCI for 12 hours per standard practice. A total of 150 patients will be randomized 1:1 to treatment of the culprit artery with IC abciximab (75 subjects) or IV abciximab (75 subjects) in addition to an infusion regimen of abciximab administered intravenously and initiated following PCI. The primary endpoint chosen to evaluate this hypothesis is infarct size as assessed on Cardiac Magnetic Resonance (CMR). Clinical outcomes will be assessed for each subject through hospital discharge and at 30 day follow-up.

Sample size: The number of patients included in this study was based on the estimation of the sample size needed to identify a statistically significant difference of the primary end-points between the two groups. The investigators estimated that 75 patients would be required in each study group to have a power of 80% to detect an absolute difference in the infarct size resolution of 15% with a two-sided alpha value of 0.05.

Conclusion: The purpose of this study is to demonstrate that an IC bolus of abciximab delivered with the ClearWay™RX catheter added to a post-PCI intravenous infusion regimen of abciximab will result in significant additional clot resolution in vivo when compared with an IV bolus of abciximab when added to a post PCI intravenous infusion regimen of abciximab. The primary endpoint chosen to evaluate this hypothesis is infarct size as assessed on CMR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (men or women) at least 18 years of age
2. STEMI: Presenting with ischemic chest discomfort > 20 minutes and <6 hours of duration suggestive of acute myocardial infarction AND ST elevation > 1 mm (> 0.1 mV) in two contiguous limb leads OR > 2 mm (> 0.2 mV) in two contiguous precordial leads
3. Must have signed the informed consent form prior to performance of study-related procedures
4. Native dominant and proximal culprit vessel 2.5 mm in diameter
5. Angiographically identifiable thrombus (presence of a filling defect within the coronary lumen surrounded by contrast medium observed in multiple projections, without calcium within the filling defect, or persistence of contrast medium within the coronary lumen)
6. Pre-PCI Thrombus score (TS) ≥ 2 (angiographically apparent thrombus that is > ½ the vessel diameter)
7. Pre-PCI TIMI flow grade of 0-2

Exclusion Criteria:

1. Previous PCI of the IRA
2. Previous myocardial infarction or coronary artery bypass grafting
3. Cardiogenic shock
4. Three vessel disease
5. Left main disease
6. Severe valvular heart disease
7. Rescue PCI (PCI following fibrinolytic administration)
8. Facilitated PCI (PCI following fibrinolytic or GP IIb/IIIa inhibition)
9. Contraindication to GP IIb/IIIa inhibitors such as excess bleeding risk or thrombocytopenia
10. Current participation in another investigational trial
11. Exclusion criteria for the MRI imaging include implanted pacemakers, defibrillators, or metallic intracranial implants, severe claustrophobia, BMI > 35 kg/m², atrial fibrillation or known not well controlled extrasystoles (bad images), or allergy to gadolinium-DTPA
12. Enrolment of patients with an estimated glomerular filtration rate < 30 ml/min/1.73 m2 should be carefully evaluated considering the gadolinium chelate-associated risk of nephrogenic systemic fibrosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Reduction in infarct size for the IC infusion group compared to the control as measured with cardiac MRI imaging | 24 months

SECONDARY OUTCOMES:
Angiographic outcomes of lesion, flow, and myocardial perfusion using established and validated Quantitative Coronary Angiographic Methodology | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Policlinico of Modena, Modena, Italy
  - Dept.of Cardiovascular Sciences,Policlinico Umberto I, Rome

REFERENCES:
- [Derived] Sardella G, Sangiorgi GM, Mancone M, Colantonio R, Donahue M, Politi L, Bucciarelli-Ducci C, Carbone I, Francone M, Ligabue G, Fiocchi F, Di Roma A, Benedetti G, Lucisano L, Stio RE, Agati L, Modena MG, Genuini I, Fedele F, Gibson M. A multicenter randomized study to evaluate intracoronary abciximab with the ClearWay catheter to improve outcomes with Lysis (IC ClearLy): trial study design and rationale. J Cardiovasc Med (Hagerstown). 2010 Jul;11(7):529-35. doi: 10.2459/JCM.0b013e3283341c1c. PMID 19918189